CLINICAL TRIAL: NCT00343824
Title: Bacterial Control in Partial Thickness Burns Using Silver-containing Wound Dressings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/224
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Burn Wounds - Partial Thickness (2nd Degree)
Keywords: Burn wounds - Silver Dressings - Bacterial Control

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- aquacel AG hydrofiber (Experimental)
  Interventions: Procedure: aquacel AG hydrofiber versus acticoat burn dressing
- Acticoat burn dressing (Experimental)
  Interventions: Procedure: aquacel AG hydrofiber versus acticoat burn dressing

INTERVENTIONS:
Procedure: aquacel AG hydrofiber versus acticoat burn dressing — Aquacel AG hydrofiber versus acticoat burn dressing will be compared.

SUMMARY:
This study is to compare the treatment with two different silver-containing wound dressings: aquacel AG hydrofiber versus acticoat burn dressing.

ELIGIBILITY:
Inclusion Criteria:

* Burn wounds with flux values, measured by Laser Doppler Imaging, corresponding with expected healing time between 7 and 21 days, flux values between 200 and 1000 (red-pink or pink-yellow-green colour)
* Wounds treated with a hydrocolloid paste prior to LDI
* Possibility to follow the complete treatment schedule until wound healing and participation on complete follow-up schedule
* Informed consent
* Partial thickness burns with TBSE < 40%

Exclusion Criteria:

* Mean flux values < 200 or > 1000
* TBSA > 40%
* Impossibility to debride necrotic skin prior to LDI measurement
* Wounds treated with any topical ointments or dressings other than hydrocolloid prior to LDI
* Not following the complete treatment schedule or missing some evaluations during the follow-up period
* Patient has any condition that seriously compromises the patient's ability to complete the study
* Patient has participated in another study using an investigational drug within the previous 30 days
* Patient has one or more medical condition(s)that in the opinion of the investigator would make the patient an inappropriate candidate for this study
* The plastic surgeon decides that surgery is necessary due to unusual circumstances
* Patient wish to decline from the study
* No informed consent
* Full thickness burns

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2006-11-01 (Actual); Primary Completion 2010-07-31 (Actual); Study Completion 2010-07-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the efficacy of both wound dressings in controlling wound bioburden over a period of 21 days | Over a period of 21 days

SECONDARY OUTCOMES:
Comparison of blood silver levels | Every week until woundhealing. In folluw-up: at 3, 6 and 12 months
Percentage of genetically-acquired resistance to silver | Once after wound closure.
Healing time comparison | Every 3 days until healing
Scar quality assessment | At 1, 3, 6 and 12 months after wound closure
Cost-effectiveness | Once after wound closure.
Health related quality of life | At 1, 3, 6 and 12 months after wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Stan Monstrey, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be